CLINICAL TRIAL: NCT00129597
Title: Effect of Ketalar to Prevent Postoperative Chronic Pain After Mastectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004.349
Record Dates: First submitted 2005-08-10; First posted 2005-08-12 (Estimated); Last update posted 2007-03-12 (Estimated); Status verified 2007-03

CONDITIONS: Pain; Breast Cancer
Keywords: Ketalar; NMDA; mastectomy; postoperative chronic pain; Chronic pain after mastectomy for breast cancer
MeSH Terms: conditions — Pain; Breast Neoplasms; Pain, Postoperative | interventions — Ketamine

INTERVENTIONS:
Drug: ketalar

SUMMARY:
Prevalence of chronic pain after mastectomy is beyond 50% 3 months after surgery. This pain is related to a sensitization of the central nervous system through N-methyl-D-asparate (NMDA) receptors. Ketalar might prevent the occurrence of chronic pain by anti-NMDA properties after mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* Mastectomy in patients 18 to 80 years old

Exclusion Criteria:

* American Society of Anesthesiology (ASA) class >= 3
* Renal, heart or hepatic failure
* Allergy to ketalar
* Psychiatric disease
* Chronic antalgic treatment

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-12

PRIMARY OUTCOMES:
To evaluate the effect of perioperative ketalar on pain intensity 3 months after a mastectomy
Pain intensity is evaluated by an appropriate questionnaire 1 and 3 months after surgery.

SECONDARY OUTCOMES:
To evaluate the incidence of chronic pain after mastectomy, the impact on life quality, and the area of hyperalgesia

CONTACTS AND LOCATIONS:
Overall Officials: Vincent PIRIOU, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France